CLINICAL TRIAL: NCT02592512
Title: Non-Invasive Ventilation With Neurally Adjusted Ventilatory Assist vs NIV Pressure Support or Pressure Control in Treatment of Patients With Acute Respiratory Insufficiency. A Prospective, Randomised, Single Blinded, Crossover Pilot Study
Brief Title: NIV-NAVA vs NIV-PS/PC in Respiratory Insufficiency
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NIV-NAVA vs NIV-PS/PC
Record Dates: First submitted 2015-10-14; First posted 2015-10-30 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Insufficiency; Acute Respiratory Insufficiency
Keywords: Hypoxia; hypercapnia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Hypercapnia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NIV-NAVA: 4 hour NIV-NAVA, followed by 4 hour NIV-PS/PC
  Interventions: Other: NIV-NAVA; Other: NIV-PS/PC
- NIV-PS/PC: 4 hour NIV-PS/PC, followed by 4 hour NIV-NAVA
  Interventions: Other: NIV-NAVA; Other: NIV-PS/PC

INTERVENTIONS:
Other: NIV-NAVA — Cross-over study where participants are randomized to start with either NIV-NAVA or NIV-PS/PC for 4 hours, followed by another 4 hours with the other arm.
Other: NIV-PS/PC — Cross-over study where participants are randomized to start with either NIV-NAVA or NIV-PS/PC for 4 hours, followed by another 4 hours with the other arm.

SUMMARY:
This study evaluates the difference between Non Invasive Ventilation with Neurally Adjusted Ventilatory Assist (NIV-NAVA) and Conventional Non Invasive Ventilation with Pressure Support (PS) or Pressure Control (PC). All the patients are ventilated in each mode for 4 hours. Afterwards they will be subjected to a semi-structured interview where they will be asked to compare the two modes. The hypothesis is that NIV-NAVA will correct patients power of Hydrogen (pH), PaCO2 og PaO2 more quickly than NIV-PS and NIV-NAVA is more comfortable for the patients.

DETAILED DESCRIPTION:
Neurally Adjusted Ventilatory Assist (NAVA) is a ventilation mode where the diaphragm is controlling the amount of ventilatory assistance proportionally through a nasogastric tube containing electrodes which are sending the electrical activities of the diaphragm (Eadi) to the ventilator.

Whereas Conventional ventilation modes like Pressure support or Pressure Control are dependent on the pressure drop or flow reversal to initiate assist delivered to the patient. This is last step of the signal chain leading to inhalation and is subject to disturbances such as intrinsic positive expiratory end pressure (PEEP), hyperinflation and leakage.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at the ICU with acute respiratory insufficiency and therefore have hypoxia(PaO2 < 7 kPa on atmospheric air) og pH < 7.35 with non-compensated hypercapnia (PaCO2 > 6.0 kPa).
* Patients, which according to the departments guidelines are required to treatment with NIV

Exclusion Criteria:

* Patients under years of 18.
* Patients without the possibility to give informed consent.
* Patients with neuromuscular or neurological disease.
* Patients with a verified or suspected head trauma.
* Patients with a acknowledged hiatus hernia.
* Patients with an active or suspected active upper GI bleeding.
* Patients which have previously been in the study.
* Patients with a suspected or verified acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU at Vejle Hospital, Denmark, with acute respiratory insufficiency.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time for normalizing of Power of Hydrogen (pH) in arterial blood gases. Normal pH frame 7.35-7.45. | 8 hours
Time for normalizing of Partial pressure of Oxygen (pO2) in arterial blood gases. Normal frame for pO2 7-14,4 (or to the usual level for the patient). | 8 hours
Time for normalizing Carbon dioxide partial pressure (pCO2) in arterial blood gases. Normal frames pCO2 4,7-6,4 (or to the usual level for the patient). | 8 hours
Electrical activity of the diaphragm (Eadi). Reduction in respiratory work assessed by Eadi (in percentage). | 8 hours

SECONDARY OUTCOMES:
Patient comfort | 24 hours
  There will be conducted a semi-interview on the subjects. They will be asked:
  If they felt any difference in breathing between the two modes. If yes, what was the difference? Which method did you prefer? And why? Do you have any comments?

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kimper-Karl, MD, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Southern Jetland, Denmark